CLINICAL TRIAL: NCT04586803
Title: Study on the Bioavailability of Three Different Prescription Processes of SHR4640 Tablets in Healthy Volunteers (Single Center, Randomized, Open, 3 Cycles, 6 Sequences)
Brief Title: Study on the Bioavailability of Three Different Prescription Processes of SHR4640 Tablets in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SHR4640-Ⅰ-109
Record Dates: First submitted 2020-09-27; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Primary Gout; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640
- B (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640
- C (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640
- D (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640
- E (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640
- F (Experimental): Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.

SUMMARY:
The primary objective of the study is to evaluate the relative bioavailability of three different prescription processes of SHR4640 tablets in healthy volunteers. The secondary objective of the study is to observe the safety of SHR4640 tablets in healthy subjects.

DETAILED DESCRIPTION:
Study Type: Interventional Enrollment: Number of Subjects: 24 Type: Anticipated

Allocation : Yes Intervention Model : Single center, randomized, open Intervention Model Description: 3 cycles, 6 sequences Masking: No Masking

Subjects were randomly divided into the group A, B, C, D, E and F. On D1, D8 and D15, six groups of subjects were respectively given A version or C version or D version of SHR4640 tablet.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntarily sign the informed consent form before the start of the activities related to this trial, and be able to understand the procedures and methods of this trial, and be willing to strictly abide by the clinical trial plan to complete this trial; 2) Aged between 18 and 45 years old (including both ends, whichever is the time of signing the informed consent form), male; 3) Body weight ≥ 50 kg, and body mass index (BMI): 19-26 kg/m2 (both ends included).

Exclusion Criteria:

* Subjects will not be allowed to enter this study if they meet any of the following criteria:

  1. General situation:
  1. Have a fertility plan within 3 months after screening to the last medication, or refuse to use medically approved contraceptive methods;
  2. Drug abusers or drug urine screening positive;
  3. Smokers (average daily smoking 5 or more) or urine Nicotin positive.
  4. The average daily alcohol intake during the first month was more than 25 g (for example, 750 mL beer, 250 mL wine or 50 mL low spirits);
  5. Anyone who had eaten grapefruit or fruit juice products within 2 days before administration, any food or drink containing caffeine (such as coffee, tea, chocolate, cola or other caffeinated carbonated drinks, etc.) and foods or drinks rich in purine food or alcohol.
  6. The researchers judged that the subjects had medical conditions that affected the absorption, distribution, metabolism and excretion of drugs or reduced compliance.

  2. Laboratory tests showed the following conditions:
  1. Those with sUA > 420 µmol / L during the screening period, or those with a previous history of hyperuricemia and / or gout;
  2. Those with estimated glomerular filtration rate (eGFR) < 90 during the screening period;
  3. Those with urolithiasis indicated or suspected by B ultrasound during the screening period;
  4. Those who were positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or syphilis antibody within one month or during the screening period.

  3. There is any history of any of the following or concomitant diseases:
  1. Any clinical history of serious illness or disease or condition that the researchers believe may affect the results of the trial, including, but not limited to, a history of circulatory, endocrine, nervous, digestive, urinary or hematological, immune, mental and metabolic diseases.
  2. People with allergies, including those who are explicitly allergic to research drugs or any ingredient in research drugs, are allergic to any food ingredient or have special requirements for diet, and are unable to follow a uniform diet;
  3. Screening those who have undergone any operation within the first 3 months, or who have not recovered after the operation, or who may have a plan for operation or hospitalization during the trial;
  4. Those who donated blood (or lost blood) within the first 3 months and donated blood (or lost blood) more than 400 mL, or received blood transfusion.

  4. Use any of the following drugs or participate in clinical trials:
  1. Screen people who have participated in clinical trials of any drug or medical device within the previous 3 months;
  2. Take any prescription drug, over-the-counter medicine, Chinese herbal medicine or dietary supplement within 2 weeks before the screening period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day1 to Day25
  Peak plasma concentration
AUC0-t | Day1 to Day25
  Area under the curve from the time of dosing. Dosing time to the last measurable (positive) concentration.
AUC0-inf(if available) | Day1 to Day25
  Area under the curve from time 0 to infinity

SECONDARY OUTCOMES:
Tmax | Day1 to Day25
  Time of maximum observed concentration
t1/2 | Day1 to Day25
  Half time
CL/F | Day1 to Day25
  apparent clearance
Vz/F | Day1 to Day25
  apparent volume of distribution
PD | Day1 to Day25
  concentration of serum urine acid

CONTACTS AND LOCATIONS:
Overall Officials: Zourong Ruan, PhD, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University

IPD SHARING:
Plan to Share IPD: No